CLINICAL TRIAL: NCT00737295
Title: Study to Investigate the Role of Ultrasound for Diagnosis of Biliary Dyskinesia
Brief Title: Ultrasound for Diagnosis of Biliary Dyskinesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution, study interest wained-so stopped.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Thomas Warren, MD, Texas Tech University Health Sciences Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TT Biliary Dyskinesia
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Biliary Dyskinesia
Keywords: Biliary; Dyskinesia; Gallbladder; Cholecystitis
MeSH Terms: conditions — Biliary Dyskinesia; Dyskinesias; Cholecystitis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- US (Experimental): There will be no experimental or control group, rather each individual will act as his/her own control.
  Interventions: Procedure: CCK Injection and Ultrasound

INTERVENTIONS:
Procedure: CCK Injection and Ultrasound — All subjects, whether they participate in this study or not, will undergo the HIDA scan as this is the accepted standard of care for diagnosing biliary dyskinesia. If a given subject agrees to participate in this study, he/she will be asked to undergo the following study procedures:
  If a pregnancy test has not already been done, a urine pregnancy test will be done for women of childbearing potential.
  An intravenous line (IV) will be inserted (if not already in place), and a standard dose of CCK (Kinevac®- 0.02 µg/kg) will then be injected according to the package insert. Ultrasound will be used to measure dimensions of the gallbladder (length, width and height) every minute for 35 minutes following injection of the CCK. This will be done by applying ultrasound jelly to the upper part of the abdomen and ultrasound probe will be used to obtain optimal images for three dimensional analysis of the subject's gallbladder.

SUMMARY:
This is a prospective, non-randomized study of 50 people with suspected biliary dyskinesia. The purpose of this study is to investigate if it is possible to use ultrasound to make a diagnosis of a condition called biliary dyskinesia. The investigators null hypothesis is that there will be no statistical difference between the proposed experimental test (Ultrasound) and the HIDA scan (a nuclear medicine hepatobiliary system scan) in the diagnosis of biliary dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects will have a suspected clinical diagnosis of biliary dyskinesia, including an ultrasound that demonstrates biliary wall thickness of < 3 mm, and no gallstones present.
2. Written informed consent document.
3. Males and Females age > 18 years

Exclusion Criteria:

1. Subjects without a suspected clinical diagnosis of biliary dyskinesia, including an ultrasound that demonstrates biliary wall thickness of > 3 mm, and/or gallstones present.
2. Pregnant or breastfeeding women
3. Subjects who do not consent to take part in the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Does ultrasound test detect contraction of gallbladder following injection of a hormone cholecystokinin (CCK), and is the degree contraction as accurate as the accepted clinical standard (the HIDA scan) for diagnosis of biliary dyskinesia. | After HIDA scan performed

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Warren, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States